CLINICAL TRIAL: NCT04184453
Title: Clinical Curative Effect Evaluation Study of Treatment of Oral Deferiprone Tablets in Aceruloplasminaemia Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Wan-Jin Chen, Professor, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRCTA,ECFAH of FMU [2019]252
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Aceruloplasminemia
Keywords: Aceruloplasminemia; Deferiprone; Pancreas MRI
MeSH Terms: conditions — Familial apoceruloplasmin deficiency

STUDY DESIGN:
Intervention Model Description: Patients who was diagnosed as aceruloplasminiaemia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferiprone treated (Experimental): Deferiprone (25 mg/kg/day) was given to the enrolled patient.
  Interventions: Drug: Deferiprone treated

INTERVENTIONS:
Drug: Deferiprone treated — Deferiprone (25 mg/kg/day) was given to the enrolled patients.
  Other Names: Clinical Curative Effect Evaluation Study of Treatment of Oral Deferiprone Tablets in Aceruloplasminaemia Patients

SUMMARY:
Aceruloplasminemia is an autosomal recessive disorder characterized by iron deposition in the brain and visceral organs. Deferiprone was used to treat aceruloplasminemia in previous study. In this study, we will assess the clinical curative effect evaluation of oral deferiprone in Chinese aceruloplasminemia patients.

DETAILED DESCRIPTION:
Diabetes is one of the most severe symptom in aceruloplasminemia. In this study, we use R2* of pancreas MRI to evaluate the effect of deferiprone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Diagnosed with aceruloplasminaemia
* Genetically confirmed diagnosis of aceruloplasminaemia

Exclusion Criteria:

* Contraindications to deferiprone therapy
* Pregnancy was excluded in women of childbearing age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-10-23 (Estimated); Study Completion 2022-11-23 (Estimated)

PRIMARY OUTCOMES:
Change of pancreas MRI | Up to 3 months
  Pancreas MRI is related to iron accumulation of pancreas
Change of glycated hemoglobin (HbA1c) | Up to 3 months
  HbA1c is a measure of long-term blood sugar control

CONTACTS AND LOCATIONS:
Overall Officials: Wanjin Chen, Principal Investigator — Department of Neurology , First Affiliated Hospital Fujian Medical University
Locations (1):
- Department of Neurology , First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China